CLINICAL TRIAL: NCT06816407
Title: The Effect of Different Doses of Prucalopride on Improving Gut Function Recovery Following Elective Colorectal Surgery: a Randomized, Double-blind Study
Brief Title: Impact of Varying Doses of Prucalopride on Improving Gut Function Recovery After Elective Colorectal Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Nouran Omar El Said, Assistant Lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HM000186
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Post-Op Complication
Keywords: pro kinetic; gut function recovery
MeSH Terms: conditions — Postoperative Complications | interventions — prucalopride; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (Placebo Comparator): Standard care
  Interventions: Other: Standard Care
- Prucalopride 2mg (Experimental): Prucalopride 2mg
  Interventions: Drug: Prucalopride 2mg; Other: Standard Care
- Prucalopride 4mg (Experimental): Prucalopride 4mg
  Interventions: Drug: Prucalopride 4mg; Other: Standard Care

INTERVENTIONS:
Drug: Prucalopride 2mg — Prucalopride 2mg taken preoperatively
  Arms: Prucalopride 2mg
Drug: Prucalopride 4mg — Prucalopride 4mg taken preoperatively
  Arms: Prucalopride 4mg
Other: Standard Care — Standard Supportive care

SUMMARY:
Postoperative ileus (POI) is a common complication after abdominal surgery, causing symptoms like nausea, vomiting, abdominal distension, and delayed passage of flatus and stool. Management remains challenging, with limited pharmacological options available. Prucalopride, a selective serotonin 5-HT4 receptor agonist, has shown promise in accelerating gastrointestinal recovery after surgery. However, the optimal timing and dosing for preventing POI remains unclear. Higher doses may provide more potent prokinetic effects in the postoperative setting. his study investigates if higher doses of prucalopride (4 mg) improve bowel function return and hospital stay in elective colorectal surgery patients compared to standard doses and placebo.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a common complication after abdominal surgery, particularly colorectal procedures, which can delay recovery and prolong hospital stay. POI is characterized by a transient cessation of coordinated bowel motility, leading to symptoms such as nausea, vomiting, abdominal distension, and delayed passage of flatus and stool. Effective management of POI remains challenging, with limited pharmacological options available. Prucalopride, a highly selective serotonin 5-HT4 receptor agonist, has shown promise in accelerating gastrointestinal recovery after surgery. However, the optimal timing and dosing of prucalopride for preventing POI remains unclear. Studies have shown dose-dependent improvements in outcomes with doses up to 4 mg daily. Higher doses may provide more potent prokinetic effects in the postoperative setting, but no studies have examined doses above 2 mg for prevention of POI in colorectal surgery. The purpose of this study is to determine if higher doses of prucalopride (4 mg) result in faster return of bowel function and shorter hospital stay compared to the standard dose (2 mg) and placebo in patients undergoing elective colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective colorectal surgery, including but not limited to colectomy, rectal resection, and sigmoid resection.

Exclusion Criteria:

* Emergency surgery
* Total colectomy
* Creation of a stoma
* Pre-existing gastrointestinal disorders
* Severe renal or hepatic impairment
* Known hypersensitivity to prucalopride.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
time to first stool | 7 days
time to tolerance of food | 7 days

SECONDARY OUTCOMES:
time to first flatus | 7 days
incidence of prolonged postoperative ileus | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Matareya Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No